CLINICAL TRIAL: NCT06877793
Title: Real-Time Diagnosis of Life-Threatening Necrotizing Soft Tissue Infections (NSTI) Using Indocyanine Green (ICG) Kinetic Modeling
Status: Recruiting | Type: Observational
Sponsor: Eric R. Henderson (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Eric R. Henderson, Associate Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: 02002719; 1R01AI184513-01 (NIH)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Necrotizing Fascitis
MeSH Terms: conditions — Fasciitis, Necrotizing | interventions — Optical Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Administration of indocyanine green (ICG) and fluorescence imaging — Patients with clinical and lab findings consistent with a diagnosis of NSTI who consent to this study will receive a one-time, weight-appropriate dose of ICG (0.2 mg/kg, in accordance with FDA-approved recommendations). Each patient will undergo fluorescence imaging immediately before and after administration of ICG.

SUMMARY:
Necrotizing soft-tissue infections (NSTIs, a.k.a. "necrotizing fasciitis" or "flesh-eating bacteria") are aggressive infections that can progress rapidly from mild symptoms to sepsis, multi-organ failure, and death. NSTI cases present with non-specific clinical, imaging, and laboratory findings, and standard-of-care techniques for NSTI diagnosis lack sensitivity and specificity, resulting in frequent misdiagnosis and delayed care, which is the single most important predictor of survival. Consequently, the cumulative mortality rate for patients with NSTIs is 20- 30%; a dire need exists for more accurate and rapid detection of NSTIs. Fluorescence-guided surgery is a nascent technology seeking to improve the recognition of anatomical structures and disease processes using fluorescent probes (fluorophores). Indocyanine green (ICG) is an FDA-approved, near-infrared fluorophore with a >60-year safety record for vascular perfusion assessment. A distinguishing histological feature of NSTIs is prominent blood vessel thrombosis in affected tissues. Leveraging these pro-thrombotic effects, our study group has demonstrated in a first-in-human study (NCT04839302) that intravenous administration of ICG and immediate fluorescence imaging reveals prominent signal deficits in NSTI-positive tissues that differentiate significantly with increased signal seen with more common-and less virulent-infections such as cellulitis. We seek now to evaluate this imaging technique on a broader scale and determine if our findings are consistent for patients affected by NSTI-causing pathogens that are not endemic to our region. This prospective, observational, multicenter clinical study will involve video-rate ICG fluorescence imaging of patients suspected of having NSTIs who present to eight tertiary, Level 1 medical centers across the United States (Aim 1). Using dynamic contrast-enhanced fluorescence imaging (DCE-FI), time profiles of ICG fluorescence intensity from different tissue pixels/regions will be extracted and parameterized to extract first-pass kinetic features. These DCE-FI features, which characterize tissue perfusion, will be evaluated alone and in combination with anonymized electronic medical record data to create a DCE-FI-based clinical decision tool and a machine- learning-based fusion (DCE FI+lab/imaging data) tool; these will be compared to identify the most accurate means of diagnosing NSTIs (Aim 2). The best-performing tool will then be evaluated-compared to current diagnostic tests-in a prospective observational clinical study of patients presenting to tertiary emergency departments with findings concerning for NSTIs (Aim 3). Based on our human study, fluorescence imaging will not delay current standard of care. To ensure data fidelity, all sites will use similar: 1) commercial fluorescence imaging systems and accessories; and 2) validated commercial fluorescence reference phantoms. Based on our early results, we have strong confidence that following rigorous testing, ICG DCE-FI will lead to an entirely new methodology for rapid identification of patients with NSTIs, which will ultimately reduce patient morbidity and improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Clinical suspicion of NSTI based on the local standard of care warranting:
* Hospital admission for observation due to suspected NSTI; and/or
* Soft tissue biopsy to rule in/out suspected NSTI; and/or
* Surgical debridement for suspected NSTI; and/or
* Specific institutional threshold criteria for triggering NSTI work-up; and
* Ability to give written informed consent.

Exclusion Criteria:

* History of allergy to ICG and/or iodine.
* Pregnant women or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED or clinic who are considered at intermediate- or high-risk for NSTI.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Determine if tissue perfusion, determined by first-pass ICG fluorescence kinetics, is reliably reduced in the setting of a necrotizing infection compared to a non-necrotizing infection. | From enrollment to the end of fluorescence imaging (about 1 day)
  We will evaluate first-pass fluorescence signal intensity changes from indocyanine green (ICG), a vascular perfusion fluorophore, in the setting of severe soft-tissue infections to determine if ICG fluorescence may be an accurate and reliable diagnostic test for differentiating life-threatening necrotizing infections from non-life-threatening non-necrotizing infections.

SECONDARY OUTCOMES:
Determine if first-pass ICG fluorescence kinetics in patients with necrotizing infections vary based on the causative bacterial species. | From enrollment to the end of imaging and lab results (about 30 days)
  In patients who had a documented necrotizing soft-tissue infection, we will compare first-pass fluorescence signal intensity changes from ICG based on the predominant causative bacterial species isolated from a patient's infection to determine if ICG signal changes vary by species.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University/Grady Memorial Hospital, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Data will only be shared in aggregate.